

## INFORMED CONSENT FORM

## PROTOCOL TITLE:

Team Science to Identify and Intervene on Metabolism- and Alcohol-Associated Liver Disease (MetALD)

## PRINCIPAL INVESTIGATOR:

Hayley Treloar Padovano, PhD

Center for Alcohol & Addiction Studies

Center for Addiction & Disease Risk Exacerbation

(401) 863-6623

hayley\_treloar@brown.edu

## DATE:

November 4, 2024

# **BROWN UNIVERSITY**



#### CONSENT FOR RESEARCH PARTICIPATION

[The SALUD Study]

You are invited to take part in a Brown University research study. Your participation is voluntary.

- RESEARCHER: The person in charge of the research study is [Dr. Hayley Padovano]. The person to talk to about being in [the SALUD study] is [Julissa, who you can call at (401) 863-XXXX], or you can talk to the person who gave you this paper.
- PURPOSE: Health matters for all people and communities. This study is testing whether
  having information about liver health helps motivate lifestyle changes. You are invited
  to think about being a part of this study because you are an adult (age 21+ years), you
  speak Spanish or English, and your lifestyle may be affecting your liver.
- PROCEDURES: Today, we will ask you about your health, take a blood sample, and ask you to respond to written questions. If the study is a good fit and you want to be in it, we will schedule two appointments, one in a few days and another about 30 days later.
  - At the first visit, your liver health will be measured with an examination called
    Fibroscan®. It is painless and does not enter your body. A team member will explain
    the exam and answer your questions now. ▲ You will talk with us again about your
    health, give a blood sample, and respond to written questions.
  - O At the end of the visit or at a convenient scheduled time, our study counselor will talk with you about your lifestyle and liver health. Our study counselor may or may not get your Fibroscan® results to share with you. See *Your Exam Results* for more information. No one will tell you what to do. Our counselor will treat you with respect and believes in your freedom to make your own choices.
  - At the second visit, you will talk with us about your health again, respond to many of the same written questions, and give a blood sample. Your counselor will also be available for a brief check-in at that appointment or by phone.
  - With your permission, your conversations with us and with your counselor may be audiotaped to make sure our team is doing their best, which means your voice will be recorded. You can say no and still be in the study.
  - For both visits, we ask you not to eat breakfast that morning, remind you of that request the day before, and provide a meal at the visit. This is because the accuracy of our blood tests depends on whether you have eaten recently, and some tests



recommend fasting for 8 hours or more. You can still be in the study if you cannot go without eating for 8 hours or more. To be in the study, however, you must agree to not eat for at least 3 hours prior to the first visit because the liver exam requires it. When you arrive at these visits, we will ask you when you last ate. If you happen to forget, your visit may need to be delayed or rescheduled.

Your Exam Results: Whether our study counselor gets your Fibroscan® results or not is decided randomly, like a coin flip. Either way, you can still request your results at the end of the study. Our study doctor who specializes in liver care reviews all scan results, and, if necessary, we will call you and send you a copy to give to your doctor. If you need help to make an appointment, find a doctor, or if you need a referral to a specialty liver clinic, we can help. A team member will answer questions **now**. ▲

*Your Blood Results:* You cannot be in this study if you have Hepatitis B or C, another preexisting liver-health condition, or our blood test results show you have Hepatitis B or C. If your blood tests are positive for Hepatitis B or C, we will let you and the RI Dept. of Health know following state law to help track disease. This is kept confidential.

#### • TIME INVOLVED:

- o Today, it will take about 1 to 1.5 hours of your time to see if you can participate.
- After today, your two study visits will each take about 3 to 4 hours. We try to schedule these in the morning because some blood tests are more accurate if you have not eaten for 8 hours or more.
- Your first conversation with our study counselor will take about 45 minutes to an hour. Your second conversation will take about 15 minutes.
- COMPENSATION: You will be paid \$30.00 for screening and \$150.00 for each visit in this study. This will add up to a total of \$330.00, if you complete all the visits, and payments will be in cash or gift cards. If you leave the study early, or if we must take you out of the study, you will only be paid for the visits you completed. We can arrange transportation at no cost to you.
- RISKS: This study has minimal risks, such as emotional discomfort from answering
  health questions or feeling pressure or coercion to participate. There are also potential
  physical risks, such as pain or discomfort associated with blood collection or fainting.
  Each time blood is collected, from 2 to 4 tablespoons of blood is drawn. It is important to
  us that you understand being in this study is your choice. No one can force you to be a
  part of this study. You can say no to any part of the study. Even if you say yes now, you
  can change your mind later. You can also take time to think it over.



- BENEFITS: Free liver screening has potential to reduce future risks of progressive liver damage and associated health risks and discomforts, which is a potential benefit. You may not directly benefit from being in this research study. If this study causes you to change your lifestyle, however, it could improve your health now or in the future.
- CONFIDENTIALITY: We try to do all we can to keep your information from being shared with people who are not a part of our research program. When we record your information or take a blood sample, we assign it a number. This number is a code to connect you to your data without using your name or other personal information. The link of your code and contact information is kept separately from your responses. Your blood samples will be stored at our Brown University laboratory until they are used for research purposes or discarded. Only our research team will have access to your data and blood samples unless you separately give your written permission for your data to be stored for future use for other research studies by qualified researchers.

To help us protect your privacy, we have a Certificate of Confidentiality (CoC). The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any requests for information that would identify you, whenever possible. The CoC cannot prevent oversight from the funding agency or Brown and will not be used to prevent disclosure of information we are mandated to report for safety.

- VOLUNTARY: You do not have to be in this study if you do not want to be. Even if you decide to be in this study, you can change your mind and stop at any time. There may also be circumstances under which we may decide to reschedule your visits or remove you from the study even if you want to continue. These include repeatedly missed appointments, apparent intoxication upon arrival to study visits, inappropriate behavior of any kind toward staff on our team, or similar circumstances. Before you say "yes" or "no" to joining this study, we want to be sure you understand the information on this paper. A team member will ask the following questions now. ▲
  - What is this study is about?
  - What is a Fibroscan®?
  - What is one thing you will be asked to do in this study?
  - Will the researchers ever tell someone you were in this study?
  - Do you have to be in this study?



| FUTURE CONTACT: Can the research team contact you in the future about research studies that may be a good fit for you? Please check "yes" or "no." You do not have to say "yes" to be this study. If you say "yes" now, you can still change your mind in the future. You can remove your name from our re-contact list at any time. | |
|---|---|
| $\square$ Yes, you may contact me in the future $\square$ No, I do not want | to be contacted |
| • CONTACT INFORMATION: If you have any questions about your participation in this study, you can call [Julissa at 401-863-XXXX or email <u>Julissa godin@brown.edu</u> ] | |
| • YOUR RIGHTS: If you have questions about your rights as a research participant, you can contact Brown University's Human Research Protection Program at 401-863-3050 or email them at <a href="mailto:IRB@Brown.edu">IRB@Brown.edu</a> . | |
| <ul> <li>CONSENT TO PARTICIPATE: Your signature below shows that you have read and<br/>understood the information in this document, and that you agree to volunteer as a<br/>research participant for this study.</li> </ul> | |
| You will be offered a copy of this form. | |
| Participant's Signature and Date / PRINTED NA | AME |



## <u>UNIVERSIDAD DE BROWN</u> CONSENTIMIENTO PARA PARTICIPAR EN INVESTIGACIÓN

El Estudio de la Salud del Hígado Versión 1, 4 de noviembre de 2024

Usted está invitado/a a participar en un estudio de investigación de la Universidad de Brown. Su participación es voluntaria.

**INVESTIGADOR:** La persona a cargo de este estudio de investigación es la Dra. Hayley Padovano. La persona con quien puede hablar sobre participar en el estudio del higado es Jacob, quien puede llamar al (401) 863-2580, o puede hablar con la persona que le entregó este documento.

**PROPÓSITO:** La salud es importante para todas las personas y comunidades. Este estudio evalúa si recibir información sobre la salud del hígado ayuda a motivar cambios en el estilo de vida. Usted está invitado/a a considerar participar en este estudio porque es un adulto (mayor de 21 años), habla español o inglés, y su estilo de vida podría estar afectando su hígado.

**PROCEDIMIENTOS:** Utilizaremos la tabla abajo para ayudar a explicar lo que le pedimos que haga en este estudio. Para la evaluación de hoy, le haremos preguntas sobre su salud, tomaremos una muestra de sangre y le pediremos que complete cuestionarios. Cada vez que se toma sangre, se extraen de 2 a 4 cucharadas. Si el estudio es adecuado para usted y desea participar, programaremos dos citas: una en unos días y otra aproximadamente 30 días después.

- Primera visita: Su salud del hígado será evaluada con un examen llamado
  Fibroscan®. Es indoloro y no entra en su cuerpo. Un miembro del equipo le
  explicará el examen y responderá a sus preguntas ahora. Hablaremos con usted
  nuevamente sobre su salud, tomaremos una muestra de sangre y le pediremos
  que responda preguntas escritas.
- Al final de la visita o en un momento programado conveniente, nuestro
  consejero del estudio hablará con usted sobre su estilo de vida y la salud de su
  hígado. Es posible que nuestro consejero reciba o no los resultados de su
  Fibroscan® para compartirlos con usted. Consulte la sección Sus resultados del
  examen para más información. Nadie le dirá qué hacer. Nuestro consejero le
  tratará con respeto y cree en su libertad para tomar sus propias decisiones.
- Segunda visita: Volveremos a hablar con usted sobre su salud, responderá muchas de las mismas preguntas escritas y tomaremos otra muestra de sangre.



Su consejero también estará disponible para un breve seguimiento en esa cita o por teléfono.

- Con su permiso, sus conversaciones con nosotros y con su consejero pueden ser grabadas en audio para asegurarnos de que nuestro equipo está haciendo su mejor trabajo, lo que significa que su voz será grabada. Puede decir que no y aun así participar en el estudio.
- Para los dos visitas, le pedimos que no desayune esa mañana. Le recordaremos esta solicitud el día anterior y le ofreceremos una comida durante la visita. Esto se debe a que la precisión de nuestros análisis de sangre depende de si ha comido recientemente, y algunas pruebas recomiendan ayunar por 8 horas o más. Aun así, puede participar en el estudio si no puede pasar 8 horas sin comer. Sin embargo, para participar, debe aceptar no comer durante al menos 3 horas antes de la primera visita porque el examen del hígado lo requiere. Cuando llegue a estas visitas, le preguntaremos cuándo comió por última vez. Si lo olvida, es posible que su visita deba ser pospuesta o reprogramada.

Sus resultados del examen: Si nuestro consejero del estudio recibe o no sus resultados del Fibroscan® se decide al azar, como un lanzamiento de moneda. De cualquier manera, puede solicitar sus resultados al final del estudio. Nuestro médico especialista en hígado revisa todos los resultados de los exámenes y, si es necesario, le llamaremos y le enviaremos una copia para que la entregue a su médico. Si necesita ayuda para programar una cita, encontrar un médico o recibir una referencia a una clínica especializada en hígado, podemos ayudarle. Un miembro del equipo responderá a sus preguntas ahora. ▲

Sus resultados de sangre: No podrá participar en este estudio si tiene Hepatitis B o C, otra condición preexistente de salud hepática, o si nuestros análisis de sangre muestran que tiene Hepatitis B o C. Si sus análisis de sangre resultan positivos para Hepatitis B o C, se lo informaremos a usted y al Departamento de Salud de Rhode Island, según la ley estatal, para ayudar a rastrear la enfermedad. Esto se mantendrá confidencial.

### **TIEMPO INVOLUCRADO:**

• Hoy, tomará aproximadamente de 1 a 1.5 horas de su tiempo para determinar si puede participar.



- Después de hoy, sus dos visitas del estudio tomarán aproximadamente de 3 a 4 horas cada una. Intentamos programarlas por la mañana porque algunos análisis de sangre son más precisos si no ha comido durante 8 horas o más.
- Su primera conversación con nuestro consejero del estudio tomará aproximadamente de 45 minutos a una hora. Su segunda conversación tomará unos 15 minutos.

## **COMPENSACIÓN:**

Usted recibirá \$30.00 por la evaluación inicial y \$150.00 por cada visita del estudio. Esto sumará un total de \$330.00 si completa todas las visitas. Los pagos se realizarán en efectivo o en tarjetas de regalo. Si abandona el estudio antes de completarlo, o si debemos retirarlo del estudio, solo recibirá el pago por las visitas que haya completado. Podemos organizar transporte sin costo para usted.

| Visita | Cuándo | Qué se hará | Cuánto tiempo tomará |
|---|---|---|---|
| Evaluación<br>inicial | Ноу | Entrevistas Cuestionarios Recolección de sangre Medidas corporales | 1 a 1.5 horas Se le pagará por las partes de la evaluación inicial que complete, incluso si el estudio no es adecuado para usted |
| Visita 1 | Esta semana o la<br>próxima | Entrevistas Cuestionarios Recolección de sangre Examen del hígado (Fibroscan®) Conversación con el consejero | 3 a 4 horas Incluye un examen del hígado (Fibroscan®) de 10 a 15 minutos. Además, tomará hasta 1 hora más, para hablar con nuestro consejero del estudio al final de la Visita 1. |
| Visita 2 | ~ 30 días después de<br>la Visita 1 | Entrevistas Cuestionarios Recolección de sangre Seguimiento con el consejero Entrevista de salida (final del estudio) | 3 to 4 horas Incluye una entrevista sobre cómo fue para usted participar en el estudio. |



RIESGOS: Este estudio tiene riesgos mínimos, como malestar emocional al responder preguntas sobre su salud o sentir presión o coerción para participar, o una violación de la confidencialidad. También existen riesgos físicos potenciales, como dolor o malestar asociado con la recolección de sangre o desmayos. Cada vez que se recolecta sangre, se extraen de 2 a 4 cucharadas. Es importante para nosotros que entienda que participar en este estudio es su elección. Su atención clínica normal fuera del estudio no se verá afectada si elige participar. Si decide finalizar su participación en el estudio, su atención clínica tampoco se verá afectada. Nadie puede obligarlo a ser parte de este estudio. Puede negarse a participar en cualquier parte del estudio. Incluso si dice que sí ahora, puede cambiar de opinión más adelante. También puede tomarse tiempo para pensarlo.

BENEFICIOS: La evaluación gratuita del hígado tiene el potencial de reducir riesgos futuros de daño hepático progresivo y los riesgos y molestias de salud asociados, lo cual es un posible beneficio. Es posible que no obtenga beneficios directos por participar en este estudio. Sin embargo, si este estudio lo lleva a cambiar su estilo de vida, podría mejorar su salud ahora o en el futuro.

CONFIDENCIALIDAD: Hacemos todo lo posible para evitar que su información sea compartida con personas que no forman parte de nuestro programa de investigación. Cuando registramos su información o tomamos una muestra de sangre, le asignamos un número. Este número es un código que conecta sus datos sin usar su nombre u otra información personal. El enlace entre su código y su información de contacto se mantiene separado de sus otras respuestas. Sus muestras de sangre se almacenarán en nuestro laboratorio de la Universidad de Brown hasta que se utilicen para fines de investigación o se descarten. Solo nuestro equipo de investigación tendrá acceso a sus datos y muestras de sangre, a menos que usted proporcione su permiso por escrito para que sus datos se almacenen para futuros estudios de investigación realizados por investigadores calificados.

Para ayudarnos a proteger su privacidad, contamos con un Certificado de Confidencialidad (CoC, por sus siglas en inglés). Los investigadores pueden usar este certificado para negarse legalmente a divulgar información que pueda identificarlo en cualquier procedimiento civil, penal, administrativo, legislativo u otro, a nivel federal, estatal o local; por ejemplo, si hay una citación judicial. Los investigadores usarán el certificado para resistir cualquier solicitud de información que lo identifique, siempre que sea posible. El CoC no puede prevenir la supervisión de la agencia financiadora o de Brown y no se usará para evitar la divulgación de información que estemos obligados a informar por razones de seguridad.



VOLUNTARIO: No tiene que participar en este estudio si no lo desea. Incluso si decide participar, puede cambiar de opinión y dejar de hacerlo en cualquier momento. También puede haber circunstancias en las que decidamos reprogramar sus visitas o excluirlo del estudio, incluso si desea continuar. Esto incluye faltar repetidamente a las citas, llegar en aparente estado de intoxicación a las visitas del estudio, comportamiento inapropiado de cualquier tipo hacia el personal de nuestro equipo u otras circunstancias similares. Antes de decir "sí" o "no" para unirse a este estudio, queremos asegurarnos de que entienda la información en este documento. Un miembro del equipo hará las siguientes preguntas ahora:

- ¿De qué se trata este estudio?
- ¿Qué es un Fibroscan®?
- ¿Cuál es una de las cosas que se le pedirá que haga en este estudio?
- ¿Los investigadores le dirán a alguien que usted estuvo en este estudio?
- ¿Tiene que participar en este estudio?

| CONTACTO FUTURO: ¿Puede el equipo de investigación contactarlo en el futuro sobre | |
|---|---|
| estudios de investigación que puedan ser adecuados para usted? Por favor, marque "sí" | |
| o "no." No tiene que decir "sí" para participar en este estudio. Si dice "sí" ahora, aún | |
| puede cambiar de opinión en el futuro. Puede eliminar su nombre de nuestra lista de | |
| recontacto en cualquier momento. | |
| ☐ Sí, pueden contactarme en el futuro | □ No, no quiero ser contactado/a |

- INFORMACIÓN DE CONTACTO: Si tiene preguntas sobre su participación en este estudio, puede llamar a Jacob al 401-863-2580 o enviar un correo electrónico a liverhealth@brown.edu.
- SUS DERECHOS: Si tiene preguntas sobre sus derechos como participante en este estudio, puede comunicarse con el Programa de Protección de Investigación Humana de la Universidad de Brown al 401-863-3050 o enviar un correo electrónico a IRB@Brown.edu.
- CONSENTIMIENTO PARA PARTICIPAR: Su firma a continuación indica que ha leído y entendido la información en este documento y que acepta participar voluntariamente como participante en este estudio.

Se le ofrecerá una copia de este formulario.



| Firma del Participante y Fecha | / | NOMBRE EN LETRA DE MOLDE |
|--------------------------------|---|--------------------------|
| Firma y Fecha del Personal | / | NOMBRE EN LETRA DE MOLDE |